CLINICAL TRIAL: NCT03323658
Title: A Phase I Dose Escalation Study of Topical Bexarotene in Women at High Risk for Breast Cancer
Brief Title: Bexarotene in Preventing Breast Cancer in Patients at High Risk for Breast Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Prevention
Other Study IDs: NCI-2017-01960; NCI-2017-01960 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); N01-CN-2012-00034; 2017-0911 (Other: M D Anderson Cancer Center); MDA2016-08-02 (Other: DCP); N01CN00034 (NIH); P30CA016672 (NIH)
Record Dates: First submitted 2017-10-26; First posted 2017-10-27 (Actual); Results first posted 2022-12-06 (Actual); Last update posted 2023-01-10 (Actual); Status verified 2022-11

CONDITIONS: Breast Atypical Ductal Hyperplasia; Breast Atypical Lobular Hyperplasia; Breast Ductal Carcinoma In Situ; Breast Lobular Carcinoma In Situ; Invasive Breast Carcinoma
MeSH Terms: conditions — Carcinoma, Intraductal, Noninfiltrating; Breast Carcinoma In Situ | interventions — Bexarotene

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Prevention (bexarotene) (Experimental): Group 1 will apply 10mg bexarotene topically to one breast QOD for 4 weeks; Group 2 will apply 10mg bexarotene topically to one breast QOD for 1 week and then daily for 3 weeks after confirmation that toxicity is at an acceptable range; Group 3 will apply 10mg bexarotene topically to one breast QOD for 1 week, then daily for 1 week, and then 20mg daily for 2 weeks after confirmation that toxicity is at an acceptable range.
  Interventions: Drug: Bexarotene; Other: Questionnaire Administration

INTERVENTIONS:
Drug: Bexarotene — Given topically
  Other Names: 3-methyl TTNEB; LGD1069; Targretin
Other: Questionnaire Administration — Ancillary studies

SUMMARY:
This phase I trial studies the side effects and best dose of bexarotene in preventing breast cancer in patients at high risk for breast cancer. Bexarotene belongs to a class of drugs that are called rexinoids, and it may reduce the incidence of breast tumors.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the recommended phase II dose of topical bexarotene 1% (weight by weight [w/w]) gel for evaluation in healthy women. (Dose Escalation Group) II. Conduct an intervention of topical 1% bexarotene gel to an unaffected breast of healthy women at high risk for breast cancer for 4 weeks at the maximum tolerated dose (MTD) as determined during the dose escalation group phase to assess bexarotene concentration in the breast tissue. (Dose Expansion Group)

SECONDARY OBJECTIVES:

I. To detect bexarotene concentration in the serum at baseline and at 4 weeks of treatment.

II. To detect bexarotene concentration in the breast tissue at 4 weeks of treatment in the dose escalation group.

III. To investigate the effects of topical bexarotene on serum biomarkers, we will determine the change from baseline in i) lipid biomarkers (total cholesterol, triglycerides, low density lipoprotein [LDL], high density lipoprotein [HDL]), ii) thyroid function biomarkers (thyroid stimulating hormone [TSH], T4, T3), iii) calcium.

EXPLORATORY OBJECTIVE:

I. To examine changes in gene expression associated with retinoid action. (Dose Expansion Group)

OUTLINE: This is a dose-escalation study.

Group 1 will apply 10mg bexarotene topically to one breast every other day (QOD) for 4 weeks; Group 2 will apply 10mg bexarotene topically to one breast every other day (QOD) for 1 week and then daily for 3 weeks after confirmation that toxicity is at an acceptable range; Group 3 will apply 10mg bexarotene topically to one breast every other day (QOD) for 1 week, then daily for 1 week, and then 20mg daily for 2 weeks after confirmation that toxicity is at an acceptable range.

After completion of study treatment, patients are followed up at 30 days.

ELIGIBILITY:
Inclusion Criteria:

* Participants must be at high risk as defined by a history of breast cancer (invasive or ductal breast carcinoma in situ [DCIS]) and be at least 5 years out from diagnosis, or lobular carcinoma in situ (LCIS), or proliferative benign breast disease such atypical ductal hyperplasia (ADH), atypical lobular hyperplasia (ALH) or genetic test confirmation of BRCA 1/2 mutation carrier or have a breast cancer risk assessment >= 1.7% in 5 years or a lifetime risk >= 20%
* No evidence of disease (in situ or invasive cancer that would normally be treated by resection) at trial entry as determined by the investigator; diagnosis of invasive cancer must be at least 5 years prior to initiation on trial
* Eastern Cooperative Oncology Group (ECOG) performance status =< 1 (Karnofsky >= 70%)
* Leukocytes >= 3,000/microliter
* Absolute neutrophil count >= 1,500/microliter
* Platelets >= 100,000/microliter
* Total bilirubin within normal institutional limits
* Aspartate aminotransferase (AST) (serum glutamic-oxaloacetic transaminase [SGOT])/alanine aminotransferase (ALT) (serum glutamate pyruvate transaminase [SGPT]) =< 1.5 x institutional upper limit of normal (ULN)
* Creatinine =< 1.5 x institutional ULN
* Hemoglobin >= 10 g/dL
* Thyroid-stimulating hormone (TSH) within normal institutional limits
* Triglycerides =< 300 mg/dl
* Total cholesterol =< 300 mg/dl
* >= 6 months from all previous breast cancer treatment (including endocrine therapy)
* Participants must have adequate accessible breast tissue as determined by the treating physician, consisting of one breast unaffected by invasive cancer, which has not been radiated; a history of benign core biopsy of this breast will be permitted
* Participants need to have had any breast imaging with a normal/benign (bi-rads 1 or 2) result within 180 days of day 0 and no further routine breast imaging planned during the course of the study (4 weeks); exception: if the mammogram result was a bi-rads 0 and the imaging work-up (ultrasound and/or magnetic resonance imaging [MRI]) result comes back normal/benign (bi-rads 1 or 2) before treatment initiation, then participant is eligible.
* For women of childbearing potential; negative pregnancy testing within 72 hours prior to or on study visit #1 (day 0) and willingness to use adequate contraception during the study intervention; OR post-menopausal defined as any one of the following 1) prior hysterectomy, 2) absence of menstrual period for 1 year in the absence of prior chemotherapy or 3) absence of menstrual period for 2 years in women with a prior history of chemotherapy exposure who were pre-menopausal prior to chemotherapy; in women of childbearing potential, effective contraception must be used for one month prior to the initiation of therapy, during therapy, and for at least one month following discontinuation of therapy; it is recommended that two reliable forms of contraception be used simultaneously; if participants are interested in enrolling and have not met the requirement for contraception, they will be seen in the clinic in 1 month for re-evaluation once they have met this requirement and ensure all other eligibility criteria is met prior to dose assignment
* Willingness to comply with all study interventions and follow-up procedures including the ability to apply the study drug to the breast
* Ability to understand and the willingness to sign a written informed consent document
* Ability to avoid exposure of the treated breast area to sunlight and artificial ultraviolet light during the use of bexarotene gel

Exclusion Criteria:

* History of allergic reactions attributed to compounds of similar chemical or biologic composition to bexarotene gel, oral or topical retinoids
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, thromboembolic disease, or psychiatric illness/social situations that would limit compliance with study requirements
* Pregnant, or had given birth, or nursed at any time during the last 12 months
* Women with a history of any cancer within the last 3 years, except for non-melanoma skin cancer; history of breast cancer must be at least > 5 years from diagnosis
* Prior bilateral breast surgery (mastectomy, segmental mastectomy, or breast augmentation surgery including breast implants or breast reductions) or combination of breast radiation and surgery involving both breasts
* Prior history or evidence of metastatic breast cancer
* Prior history of histologically confirmed bilateral invasive breast cancer
* Current use or < 6 months since use of selective estrogen receptor modulator (SERMS) or aromatase inhibitors or any other investigational treatment for breast cancer prevention or therapy
* Skin lesions that disrupt the stratum corneum (e.g., eczema, ulceration) or any breakdown of the skin
* Current use of a retinol containing agent or any retinoid analogue drug within the last 30 days
* Dietary vitamin A intake >= 5,000 IU/day (as determined by dietary supplementation)
* Treatment with any investigational drug or investigational biologic within 30 days of initiating study treatment or during the study
* History of human immunodeficiency virus (HIV) or active hepatitis C

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2018-06-15 (Actual); Primary Completion 2021-08-03 (Actual); Study Completion 2022-03-25 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Parijatham (Priya) S Thomas, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Women at high risk for breast cancer were recruited for the trial at the Cancer Prevention Center at MD Anderson Cancer Center.
Pre-assignment Details: 41 participants were consented, 17 were not randomized due to (1 )Dose escalation phase closed and (16) were not eligible.
Groups:
- Dose Level 1; Expansion Cohort: Bexarotene 1 % gel 10 mg every other day
- Dose Level 2: Bexarotene 1 % gel 10 mg daily
Period: Overall Study
Arm/Group | Dose Level 1 | Dose Level 2 | Expansion Cohort
Started | 10 | 4 | 10
Completed | 10 | 3 | 10
Not Completed | 0 | 1 | 0
Not completed — Adverse Event | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Dose Level 1 | Dose Level 2 | Expansion Cohort | Total
Number analyzed (Participants) | 10 | 4 | 10 | 24
Age, Customized [Count of Participants; unit: Participants]
  40-49 years | 2 | 0 | 1 | 3
  50-59 years | 3 | 0 | 6 | 9
  60-69 years | 5 | 3 | 2 | 10
  70 and over years | 0 | 1 | 1 | 2
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 4 | 10 | 24
  Male | 0 | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 10 | 4 | 9 | 23
  Unknown or Not Reported | 0 | 0 | 1 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 2 | 1 | 1 | 4
  White | 8 | 3 | 8 | 19
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 1 | 1
Region of Enrollment [Number; unit: participants]
  United States | 10 | 4 | 10 | 24
Menopause [Count of Participants; unit: Participants]
  Pre-Menopausal | 2 | 0 | 3 | 5
  Post-Menopausal | 8 | 4 | 7 | 19

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Incidence of Adverse Events (Dose Limiting Toxicities)
Description: Dose Limiting Toxicity (DLT) is defined as a grade 2 skin adverse event that persists for at least 6 days or any grade 3 or greater adverse event possibly, probably, or definitely related to the study drug. In addition, a DLT will be a grade 2 skin adverse event that recurs and persists for at least 3 days.
Time Frame: 4 weeks of treatment, Up to 30 days after completion of study drug for AE assessments
Measure: Count of Participants; unit: Participants
Arm/Group | Dose Level 1 | Dose Level 2 | Expansion Cohort
Number analyzed (Participants) | 10 | 4 | 10
Participants
  Maculopapular rash with pruritus at application site | 0 | 1 | 1
  Erythema/redness at application site | 0 | 1 | 0

2. Secondary Outcome: Number of Participants With Changes in Markers of Systemic Toxicity
Description: Serum biomarkers to be tested will be total cholesterol, triglycerides, low-density lipoprotein, high-density lipoprotein, thyroid-stimulating hormone, T4, T3, and calcium. Will be summarized using mean, standard deviation and median (range) for continuous variables at each time point. Wilcoxon rank-sum test may be used to examine the difference of continuous variables between participants' characteristics groups. Will be plotted as functions of time (baseline, week 1, week 2, and week 4). Linear mixed effect model will be applied to model the biomarker change over time for all participants. Appropriate transformation and regression model will be used to ensure the model fit.
Time Frame: Baseline up to 28 days
Measure: Count of Participants; unit: Participants
Groups:
- Dose Level 1; Expansion Cohort: Bexarotene 1 % gel 10 mg QOD
- Dose Level 2: Bexarotene 1 % gel 10 mg QD
Arm/Group | Dose Level 1 | Dose Level 2 | Expansion Cohort
Number analyzed (Participants) | 10 | 4 | 10
Participants | 0 | 0 | 1

3. Secondary Outcome: Number of Participants With Trace Level of Bexarotene Concentration in Plasma Detected
Description: Plasma concentrations of bexarotene were evaluated in all participants at baseline and at end of study. Plasma samples: ND = Not detected (below the quantitation limit of 0.5 ng/mL) TDL = Trace levels detected (below the LOQ of 0.5ng/mL; estimated value)
Time Frame: baseline and end of treatment, up to 4 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Dose Level 1 | Dose Level 2 | Expansion Cohort
Number analyzed (Participants) | 10 | 4 | 10
Participants
  Plasma Baseline Visit | 0 | 0 | 0
  Plasma End of Treatment Visit | 0 | 0 | 2

4. Secondary Outcome: Number of Participants With Bexarotene Concentration in Tissue
Description: Breast tissue concentrations were available only in those women who underwent breast biopsies. Tissue samples: Not detected (below the quantitation limit of 2.5 ng/g for a 10mg sample) and Trace levels detected (below the LOQ of 2.5ng/g; estimated value).
Time Frame: end of treatment, up to 4 weeks
Population: 1 participant was to analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | Dose Level 1 | Dose Level 2 | Expansion Cohort
Number analyzed (Participants) | 5 | 1 | 9
Participants
  Non Detected | 1 | 0 | 4
  Trace Levels Detected | 1 | 0 | 2
  Quantitation limit of 2.6-10 ng/g | 1 | 0 | 1
  Quantitation limit of 11-20 ng/g | 1 | 1 | 1
  Quantitation limit of 21-30 ng/g | 1 | 0 | 0
  Quantitation limit of >30 ng/g | 0 | 0 | 1

5. Other Pre Specified Outcome: Tissue Markers
Description: One of the four cores collected from the core biopsies from baseline (in dose expansion cohort only) and post treatment (all dose expansion cohort participants and optional for dose escalation group) will be formalin-fixed and paraffin embedded (FFPE) for histological analysis. One of the four cores collected from the core biopsies from baseline and post treatment will be placed in RNALater and utilized for gene expression of ribonucleic acid (RNA) biomarkers. Gene expression will be performed.
Time Frame: baseline, 15, and Day 28 visits
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: 4 weeks of treatment, Up to 30 days after completion of study drug for AE assessments
Arm/Group | Dose Level 1 | Dose Level 2 | Expansion Cohort
All-Cause Mortality (participants affected / at risk) | 0/10 | 0/4 | 0/10
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/4 | 0/10
Other Adverse Events (participants affected / at risk) | 9/10 | 4/4 | 10/10
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Dose Level 1 (N=10) | Dose Level 2 (N=4) | Expansion Cohort (N=10)
Motion Sickness (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
General Disorders and Administration Site Conditions-Other, Specify (General disorders) | 1 (1) | 0 (0) | 0 (0) — Rash/papulopustular(w/o pustules) at site application
General Disorders and Administration Site Conditions-Other, Specify (General disorders) | 3 (3) | 0 (0) | 0 (0) — Burning sensation on rash at site application
General Disorders and Administration Site Conditions-Other, Specify (General disorders) | 3 (3) | 2 (2) | 3 (3) — Rash/maculo/papular at site application
General Disorders and Administration Site Conditions-Other, Specify (General disorders) | 8 (11) | 1 (2) | 7 (9) — Itching/pruritis at site application
General Disorders and Administration Site Conditions-Other, Specify (General disorders) | 0 (0) | 1 (4) | 0 (0) — Maculopapular rash with intermittent pruritus at site application
General Disorders and Administration Site Conditions-Other, Specify (General disorders) | 1 (4) | 1 (1) | 2 (2) — Erythema/redness (non-painful) at application site
Tired(Fatigue) (General disorders) | 1 (1) | 1 (1) | 0 (0)
General Disorders and Administration Site Conditions-Other, Specify (General disorders) | 1 (1) | 0 (0) | 0 (0) — Sun burn/rash macular without papules (includes itching) at application site
General Disorders and Administration Site Conditions-Other, Specify (General disorders) | 1 (1) | 0 (0) | 0 (0) — Tingling sensation at site application
Tongue Swelling/soreness (General disorders) | 1 (1) | 0 (0) | 0 (0)
General Disorders and Administration Site Conditions-Other, Specify (General disorders) | 2 (3) | 0 (0) | 0 (0) — Fine maculopapular rash at application site
General Disorders and Administration Site Conditions-Other, Specify (General disorders) | 0 (0) | 1 (1) | 0 (0) — Dryness at application site
General Disorders and Administration Site Conditions-Other, Specify (General disorders) | 1 (1) | 0 (0) | 0 (0) — Rash (papular) at application site (20%)
General Disorders and Administration Site Conditions-Other, Specify (General disorders) | 0 (0) | 1 (1) | 0 (0) — Redness with some mild intermittent rash over approximately 60% of left chest including superior aspect of left breast to below left clavicle "entire application site"
General Disorders and Administration Site Conditions-Other, Specify (General disorders) | 0 (0) | 1 (1) | 0 (0) — Redness with faint rash over left chest including superior aspect of left breast
General Disorders and Administration Site Conditions-Other, Specify (General disorders) | 0 (0) | 0 (0) | 1 (1) — Rash (painless erythema) over 50-75% of application area
General Disorders and Administration Site Conditions-Other, Specify (General disorders) | 0 (0) | 0 (0) | 1 (1) — Rash (painless erythema) less than 50% of application area
General Disorders and Administration Site Conditions-Other, Specify (General disorders) | 0 (0) | 0 (0) | 1 (1) — Occasional warm sensation inside upper portion of right breast on some days of gel application
General Disorders and Administration Site Conditions-Other, Specify (General disorders) | 0 (0) | 0 (0) | 1 (1) — Small red bumps/dots on the left breast at application site.
General Disorders and Administration Site Conditions-Other, Specify (General disorders) | 0 (0) | 0 (0) | 1 (1) — Rash Acneiform, single red raised spot, with few small scattered spots at application site
General Disorders and Administration Site Conditions-Other, Specify (General disorders) | 0 (0) | 0 (0) | 1 (1) — Raw Blister-like area on left breast at site of steri-strip from biopsy procedure
Dermatitis (blistering) (Immune system disorders) | 0 (0) | 1 (1) | 0 (0)
Allergic reaction, small itchy lump on right arm at allergy shot injection site (Immune system disorders) | 1 (1) | 0 (0) | 0 (0)
COVID-19 (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Absolute neutrophil count decreased (Investigations) | 0 (0) | 0 (0) | 1 (1)
Hypertriglyceridemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 1 (1) | 0 (0) | 1 (1)
Dysgeusia (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) — Tin (metallic) taste in mouth approximately 2 hours after applying gel
Depression (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
Sleep disturbance/insomnia (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
Breast Tenderness (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0)
Reproductive System and Breast Disorders-Other, Specify (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0) — Vaginal itchiness
Reproductive System and Breast Disorders-Other, Specify (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1) — Heaviness (fullness) in right breast
Cough/Coughing (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 0 (0)
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
General Disorders and Administration Site Conditions-Other, Specify (General disorders) | 1 (1) | 0 (0) | 0 (0) — Rash/papulopustular (w/o pustules) of sternum and not at site application
General Disorders and Administration Site Conditions-Other, Specify (General disorders) | 1 (1) | 0 (0) | 0 (0) — Itching of upper outer quadrant of left breast, not at application site
Pain of Skin (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) — Burning sensation on skin underneath and on the side of breast (not at application site)
Rash Maculopapular (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) — Maculopapular rash with intermittent pruritus (not at site application)
Rash Maculopapular (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) — Maculopapular rash on sides of right breast (not site of application)
Skin and Subcutaneous Tissue Disorders - Other, Specify (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) — Erythema/redness (non-painful) along bra wire line (not at application site)
Skin and Subcutaneous Tissue Disorders- Other, Specify (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) — Singular pale red patch, same location above bilateral breast that may be related to the use of the tank top (not at application site)
Skin and Subcutaneous Tissue Disorders - Other, Specify (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) — Redness/burning irritation on skin from pre-biopsy cleansing scrub
Pruritus (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0) | 0 (0)
General Disorders and Administration Site Conditions-Other, Specify (General disorders) | 0 (0) | 0 (0) | 1 (1) — Erythema (intermittent) small reddened area at application site
General Disorders and Administration Site Conditions-Other, Specify (General disorders) | 0 (0) | 0 (0) | 1 (1) — Erythema (redness) on left breast at site of steri-strips from biopsy procedure
Skin and Subcutaneous Tissue Disorders - Other, Specify (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) — Burning sensation on skin underneath and on the side of breast (not at application site)
General Disorders and Administration Site Conditions-Other, Specify (General disorders) | 0 (0) | 0 (0) | 1 (1) — Rash on upper medial portion of right breast at the application site
Skin and Subcutaneous Tissue Disorders - Other, Specify (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) — Rash papulopustular (without pustules) of sternum and not at application site

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-04-27): https://cdn.clinicaltrials.gov/large-docs/58/NCT03323658/Prot_SAP_000.pdf